CLINICAL TRIAL: NCT00320008
Title: Intensified Multifactorial Intervention in Patients With Type 2 Diabetes and Microalbuminuria
Acronym: Steno-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peter Gæde (Other)
Responsible Party: Sponsor-Investigator, Peter Gæde, Associate Professor, Steno Diabetes Center Copenhagen
Organization: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA92071gm
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Treatment Arm (Active Comparator): This arm will at any time during the active intervention period follow treatment guidelines by the Danish Medical Association for the treatment of type 2 diabetes.
  Interventions: Behavioral: Diet; Behavioral: Exercise; Behavioral: Stop smoking; Drug: Glucose lowering therapy; Drug: Blood pressure lowering therapy; Drug: Lipid lowering therapy
- Intensive Treatment Arm (Experimental): This arm will during the active intervention period be treated according to intensified multiple risk factor intervention following strict guidelines set out by the study protocol.
  Interventions: Behavioral: Diet; Behavioral: Exercise; Behavioral: Stop smoking; Drug: Glucose lowering therapy; Drug: Blood pressure lowering therapy; Drug: Lipid lowering therapy

INTERVENTIONS:
Behavioral: Diet
Behavioral: Exercise
Behavioral: Stop smoking
Drug: Glucose lowering therapy
Drug: Blood pressure lowering therapy
Drug: Lipid lowering therapy

SUMMARY:
The purpose of this study is to determine whether intensified multifactorial intervention comprising both behaviour modification and polypharmacy can reduce the risk for late diabetic complications compared to standard treatment in patients with type 2 diabetes and microalbuminuria.

DETAILED DESCRIPTION:
The overall description of the Steno-2 Study is stated in four protocols approved by the regulatory authorities in Denmark. The protocol identification numbers are KA 92071gm (4 years intervention ), KA-99035g (8 years intervention ), KA-99035-GS (13 years follow-up since intervention start) and H-KA-99035-GS (21 year follow-up since intervention start).

The aim of the study was to determine whether intensified multifactorial intervention comprising both behaviour modification and polypharmacy can reduce the risk for late diabetic complications compared to standard treatment in patients with type 2 diabetes and microalbuminuria. The primary end point after four years of intervention was to progression to diabetic nephropathy with other microvascular complications as secondary end points. The primary end point after eight years of intervention was a composite CVD endpoint with microvascular complications as secondary end points.

The interventional part of the study was ended in December 2001 after a total of eight years of intervention. From that time on, all patients were followed in a post-trial study. Also, during post-trial period all patients in both original treatment arms received similar treatment resembling the treatment given in the original intensive arm of the study. The aim of the post-trial follow-up was to investigate the effect of intensified multifactorial intervention on i) mortality and ii) years of life gained, respectively, with such an interventional approach.

Endpoints in the two parts of the post-trial follow-up:

Part one at 13 years since start of intervention:

Primary endpoint: Total mortality. Secondary endpoints: Cardiovascular endpoints as defined previously; Microvascular disease.

Part two at 21 years since start of intervention:

Primary endpoint: Difference in median time to 50% mortality in each of the two original treatment groups Secondary endpoints: Cardiovascular endpoints as defined previously; Recurrent cardiovascular events; Microvascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Microalbuminuria

Exclusion Criteria:

* Stimulated serum C-peptide concentration less than 600 pmol/L
* Pancreatic insufficiency or diabetes secondary to pancreatitis
* Alcohol abuse
* Non-diabetic kidney disease
* Life-threatening disease with death probable within 4 years of study start

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 1992-01; Primary Completion 2001-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diabetic nephropathy | Four years
Combined cardiovascular endpoint | Eight years
Total mortality | 13 years
Years of life years gained | 21 years

SECONDARY OUTCOMES:
All cause mortality | 22 years
Cardiovascular disease mortality | 22 years
Stroke | 22 years
Myocardial infarction | 22 years
Coronary interventions | 22 years
Amputations | 22 years
Vascular surgery | 22 years
Diabetic retinopathy | 22 years
Diabetic nephropathy | 22 years
Diabetic neuropathy | 22 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gaede, Professor, Study Director — Slagelse Hospital
Locations (1):
- Slagelse Hospital, Slagelse, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gaede P, Vedel P, Parving HH, Pedersen O. Intensified multifactorial intervention in patients with type 2 diabetes mellitus and microalbuminuria: the Steno type 2 randomised study. Lancet. 1999 Feb 20;353(9153):617-22. doi: 10.1016/S0140-6736(98)07368-1. PMID 10030326
- [Result] Gaede P, Vedel P, Larsen N, Jensen GV, Parving HH, Pedersen O. Multifactorial intervention and cardiovascular disease in patients with type 2 diabetes. N Engl J Med. 2003 Jan 30;348(5):383-93. doi: 10.1056/NEJMoa021778. PMID 12556541
- [Result] Gaede P, Lund-Andersen H, Parving HH, Pedersen O. Effect of a multifactorial intervention on mortality in type 2 diabetes. N Engl J Med. 2008 Feb 7;358(6):580-91. doi: 10.1056/NEJMoa0706245. PMID 18256393
- [Result] Gaede J, Oellgaard J, Ibsen R, Gaede P, Nortoft E, Parving HH, Kjellberg J, Pedersen O. A cost analysis of intensified vs conventional multifactorial therapy in individuals with type 2 diabetes: a post hoc analysis of the Steno-2 study. Diabetologia. 2019 Jan;62(1):147-155. doi: 10.1007/s00125-018-4739-3. Epub 2018 Oct 6. PMID 30293113
- [Result] Oellgaard J, Gaede P, Persson F, Rossing P, Parving HH, Pedersen O. Application of urinary proteomics as possible risk predictor of renal and cardiovascular complications in patients with type 2-diabetes and microalbuminuria. J Diabetes Complications. 2018 Dec;32(12):1133-1140. doi: 10.1016/j.jdiacomp.2018.09.012. Epub 2018 Sep 24. PMID 30282584
- [Result] Kjaer LK, Oellgaard J, Henriksen T, Gaede P, Pedersen O, Poulsen HE. Indicator of RNA oxidation in urine for the prediction of mortality in patients with type 2 diabetes and microalbuminuria: A post-hoc analysis of the Steno-2 trial. Free Radic Biol Med. 2018 Dec;129:247-255. doi: 10.1016/j.freeradbiomed.2018.09.030. Epub 2018 Sep 21. PMID 30244028
- [Result] Oellgaard J, Gaede P, Rossing P, Persson F, Parving HH, Pedersen O. Intensified multifactorial intervention in type 2 diabetics with microalbuminuria leads to long-term renal benefits. Kidney Int. 2017 Apr;91(4):982-988. doi: 10.1016/j.kint.2016.11.023. Epub 2017 Feb 7. PMID 28187983
- [Result] Oellgaard J, Gaede P, Rossing P, Rorth R, Kober L, Parving HH, Pedersen O. Reduced risk of heart failure with intensified multifactorial intervention in individuals with type 2 diabetes and microalbuminuria: 21 years of follow-up in the randomised Steno-2 study. Diabetologia. 2018 Aug;61(8):1724-1733. doi: 10.1007/s00125-018-4642-y. Epub 2018 May 30. PMID 29850922
- [Result] Gaede P, Oellgaard J, Carstensen B, Rossing P, Lund-Andersen H, Parving HH, Pedersen O. Years of life gained by multifactorial intervention in patients with type 2 diabetes mellitus and microalbuminuria: 21 years follow-up on the Steno-2 randomised trial. Diabetologia. 2016 Nov;59(11):2298-2307. doi: 10.1007/s00125-016-4065-6. Epub 2016 Aug 16. PMID 27531506
- [Derived] Cashmore BA, Cooper TE, Evangelidis NM, Green SC, Lopez-Vargas P, Tunnicliffe DJ. Education programmes for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 Aug 22;8(8):CD007374. doi: 10.1002/14651858.CD007374.pub3. PMID 39171639
- [Derived] Do DV, Han G, Abariga SA, Sleilati G, Vedula SS, Hawkins BS. Blood pressure control for diabetic retinopathy. Cochrane Database Syst Rev. 2023 Mar 28;3(3):CD006127. doi: 10.1002/14651858.CD006127.pub3. PMID 36975019
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Gaede P, Oellgaard J, Kruuse C, Rossing P, Parving HH, Pedersen O. Beneficial impact of intensified multifactorial intervention on risk of stroke: outcome of 21 years of follow-up in the randomised Steno-2 Study. Diabetologia. 2019 Sep;62(9):1575-1580. doi: 10.1007/s00125-019-4920-3. Epub 2019 Jun 1. PMID 31154479
- [Derived] Gaede P, Valentine WJ, Palmer AJ, Tucker DM, Lammert M, Parving HH, Pedersen O. Cost-effectiveness of intensified versus conventional multifactorial intervention in type 2 diabetes: results and projections from the Steno-2 study. Diabetes Care. 2008 Aug;31(8):1510-5. doi: 10.2337/dc07-2452. Epub 2008 Apr 28. PMID 18443195